CLINICAL TRIAL: NCT03968549
Title: Study of the Importance of Intestinal Microbiota in Patients With Heart Failure - Randomized, Double-blind Study
Brief Title: Probiotics and Inflammatory Status in Patients With Heart Failure
Acronym: PROBHF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Fernando Bacal, Director of Heart Transplant Unit, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROBHF
Record Dates: First submitted 2018-11-01; First posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Heart Failure
Keywords: Probiotics; Inflammation; Heart failure; Intestinal microbiota
MeSH Terms: conditions — Heart Failure; Inflammation | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): These patients will receive capsules containing vegetable oil and corn starch
  Interventions: Other: Placebo
- Probiotic (Active Comparator): These patients will receive capsules containing Lactobacillus acidophilus
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Those patients in group Probiotic will receive the capsules containing Lactobacillus acidophilus and will need to take one of it everyday during the study.
  Arms: Probiotic
Other: Placebo — Those patients in group Placebo will receive the capsules containing vegetable oil and corn starch and will need to take one of it everyday during the study.
  Arms: Placebo

SUMMARY:
Cachexia is a very common condition in patients with advanced heart failure (HF) and is considered a predictor of mortality. Studies have been carried out in an attempt to discover the mechanisms that leads to cachexia in order to improve the therapies and the survival of these patients. Some of these studies give the hypothesis that the gastrointestinal tract, more precisely the intestine, can collaborate with cachexia. Some of these studies suggest that, the intestinal mucosa, due to hypoperfusion, becomes more permeable to some substances, as like endotoxins, being the lipopolysaccharide (LPS) one of them. The circulating LPS can stimulate the increase of tumor necrosis alpha (TNF-alpha) further increasing the inflammation and, consequently, contributing to the worsening of prognosis. The intestinal microbiota is also affected by hypoperfusion, contributing with increase of permeability. As known, probiotics can help to maintain or recover the microbiota and maintain a healthy intestinal barrier. In view of the importance of microbiota to inflammation in the prognosis of the patients and the performance of microbiota in maintenance of intestinal barrier, this study has as primary objective to verify the influence of supplementation of the probiotic Lactobacillus acidophilus (LA) in the lowering of serum levels of TNF-alpha in the patients with HF.

DETAILED DESCRIPTION:
The present study will be a clinical trial compounded by two parallel arms, randomized, double-blind (researcher-patient), placebo-controlled, with patients with heart failure (HF), functional class according the New York Heart Association (NYHA) III and IV. It will be included 58 patients, 29 will receive probiotics and 29 will receive placebo. These patients will be accompanied during 6 months and should take one capsule every day during the study. In the beginning of the study and at the end, venous blood sample will be collected of each patient for laboratory measurement of TNF alpha, interleukins 1,6 and 10, LPS, B-type natriuretic peptide (BNP) and C-reactive protein (CRP). To establish the normality pattern of these markers studied, a control group, with healthy individuals, will be performed.An anthropometric evaluation will be performed with measurements of weigh, height, arm circumference, triceps skin fold. According to nutritional status, it will be calculated the caloric and protein needs of each patient and, to monitor the consumption, in each consult will be applied the 24-hour food recall and calculated the consumption from it. In order to measure the appetite of the patients, in each consult, an appetite questionnaire will be applied. To statistical analysis, the test of Kolmogorov-Smirnov will be used to assess whether the distribution is normal for the quantitative variables. If the variable follows normal distribution, it will be described as mean and standard deviation, otherwise, it will be described as median and interquartile range. The groups will be compared using t-Student or Mann-Whitney tests. The categorical variables will be presented descriptively with absolute and relative frequencies. The association between categorical variables will be analyzed with chi square test or Fisher exact test or likelihood ratio test. For the repeated measures, will be used the ANOVA test or Friedman test and Wilcoxon signs. The analyzes will be performed according to the intent-to-treat principle and the two-tailed tests. The value of p<0,5 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart failure NYHA functional class III and IV;
* Medications optimized for at least 2 months;
* No hospitalizations for HF decompensated or acute myocardial infarction in the last 30 days;
* Have signed the Free and Informed Consent Form

Exclusion Criteria:

* Do not accept to participate in the study or do not signed the Free and Informed Consent Form
* Have used antibiotics and/or corticosteroids in the last 30 days;
* Clinical conditions that can affect the inflammatory profile such as inflammatory bowel disease, arthrosis, among others;
* Be pregnant;
* Have been submitted to a cardiac surgery in the last 6 months or other surgery in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Effects of probiotics in serum levels of TNF-alpha | six months
  Probiotics should improve serum levels of tumor necrosis alpha (TNF-alpha)

SECONDARY OUTCOMES:
Effects of probiotics in serum levels of lipopolysaccharide LPS (ng/mL) | six months
  Probiotics should improve serum levels of LPS (ng/mL)
Effects of probiotics in serum levels of interleukin 1 (IL 1) (pg/mL) | six months
  Probiotics should improve serum levels of IL 1 (pg/mL)
Effects of probiotics in serum level of interleukin 6 (IL 6) (pg/mL) | six months
  Probiotics should improve serum levels of IL 6 (pg/mL)
Effects of probiotics in serum levels of interleukin 10 (IL 10)(pg/mL) | six months
  Probiotics should improve serum levels of IL 10 (pg/mL)
Effects of probiotics in serum levels of B-type natriuretic peptide (BNP) (pg/mL) | six months
  Probiotics should improve serum levels of BNP (pg/mL)
Effects of probiotics in serum levels of C-reactive protein (CRP) (mg/L) | six months
  Probiotics should improve serum levels of CRP (mg/L)
Effects of probiotics in appetite | six months
  Probiotics should improve the appetite

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Bacal, MD PhD, Principal Investigator — Heart Institute (InCor), University of Sao Paulo, Medical School
Locations (1):
- Fernando Bacal, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No